CLINICAL TRIAL: NCT00324870
Title: Phase I/II Study of Suberoylanilide Hydroxamic Acid (SAHA) in Combination With the VEGF Inhibitor Bevacizumab in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Vorinostat and Bevacizumab in Treating Patients With Unresectable or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00093; NCI-2009-00093 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NA 00001107; NCI-6884; JHOC-J0570; CDR0000467800; 6884; JHOC-00001107; J0570; IRB #NA 00001107, SKCCC J0570 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 6884 (Other: CTEP); P30CA006973 (NIH); U01CA062491 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2013-10

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Vorinostat; Bevacizumab

ARMS (1):
- Arm I (Experimental): Phase I: Patients receive oral SAHA twice daily on days 1-14 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.
  Phase II: Patients receive SAHA at the MTD determined in phase I and bevacizumab as in phase I.
  Interventions: Drug: vorinostat; Drug: bevacizumab

INTERVENTIONS:
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Drug: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF

SUMMARY:
This phase I/II trial is studying the side effects and best dose of vorinostat when given together with bevacizumab and to see how well they work in treating patients with unresectable or metastatic kidney cancer. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of kidney cancer by blocking blood flow to the tumor. Giving vorinostat together with bevacizumab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety and tolerability of vorinostat (SAHA) in combination with bevacizumab in patients with unresectable or metastatic renal cell carcinoma. (Phase I) II. Determine the recommended dosing in patients treated with this regimen. (Phase I) III. Determine the proportion of patients who are progression-free at 6 months after receiving this regimen. (Phase II) IV. Determine the clinical response rate in patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. Determine the toxicity of this regimen in these patients. (Phase II) II. Determine time to progression and duration of progression-free and overall survival in patients treated with this regimen. (Phase II) III. Determine the pharmacodynamic effects in peripheral blood mononuclear cells and tumors before and after treatment with this regimen in these patients. (Phase II) IV. Determine the antiproliferative and apoptotic effects of this regimen in these patients. (Phase II) V. Determine the antiangiogenic effects of this regimen in these patients. (Phase II) VI. Determine the modulation of tumor metabolism and tumor blood flow in patients treated with this regimen. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of vorinostat (SAHA) followed by a phase II study.

PHASE I: Patients receive oral SAHA twice daily on days 1-14 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.

PHASE II: Patients receive SAHA at the MTD determined in phase I and bevacizumab as in phase I.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* No known CNS metastasis
* ECOG performance status 0-2
* Life expectancy > 6 months
* LVEF ≥ 45%
* Absolute neutrophil count ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 50 mL/min
* PT/INR ≤ 1.5
* Urine protein < 1+ by urinalysis OR < 1 g by 24-hour urine collection
* Not pregnant
* No nursing during and for 6 months after completion of study treatment
* Negative pregnancy test
* Fertile patients must use effective contraception for 2 weeks prior, during, and for 6 months after completion of study treatment
* No other currently active malignancy defined as > 30% risk of relapse upon completion of anticancer therapy, except nonmelanoma skin cancer
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to vorinostat (SAHA)
* No hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* No evidence of bleeding diathesis or coagulopathy
* No active bleeding or pathological conditions that carry high risk of bleeding (i.e., tumor involving major vessels or known varices)
* No ongoing, active infection
* No New York Heart Association class II-IV congestive heart failure
* No angina pectoris requiring nitrate therapy
* No cardiac arrhythmia
* No myocardial infarction within the past 6 months
* No history of cerebrovascular accident within the past 6 months
* No uncontrolled hypertension (defined as systolic blood pressure (BP) > 160 mm Hg and/or diastolic BP > 90 mm Hg on medication)
* No history of peripheral vascular disease
* No psychiatric illness or social situation that would preclude study compliance
* No other uncontrolled illness
* No serious nonhealing wound, ulcer, or bone fracture
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No significant traumatic injury in the past 28 days
* At least 4 weeks since prior major surgery or open biopsy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* More than 4 weeks since prior radiotherapy
* At least 2 weeks since prior tyrosine kinase inhibitor
* Prior palliative radiotherapy to metastatic lesions allowed provided ≥ 1 measurable and/or evaluable lesion has not been irradiated
* No more than 2 prior systemic treatments for metastatic disease, including immunotherapy, receptor tyrosine kinase inhibitor therapy, chemotherapy, or investigational therapy
* No prior therapy with bevacizumab, vascular endothelial growth factor-trap, or histone deacetylase inhibitors, including valproic acid
* No core biopsy within 1 week prior to day 1 of study treatment
* No planned major surgery during study treatment
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* Concurrent stable-dose prophylactic anticoagulation (i.e., warfarin or low molecular weight heparin) allowed provided requirements for INR are met
* Histologically confirmed renal cell carcinoma, clear cell component, unresectable or metastatic disease (patients with a primary tumor in place who are eligible for surgery are strongly encouraged to undergo a nephrectomy prior to study entry to increase potential survival)
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques OR ≥ 10 mm with spiral CT scan
* The following histologies are not allowed:

  * Papillary, sarcomatoid carcinoma
  * Chromophobe carcinoma
  * Oncocytoma
  * Collecting duct tumor
  * Transitional cell carcinoma
* WBC ≥ 3,000/mm^3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-02; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Carducci, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (3):
- United States (3):
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Peninsula Oncology and Hematology PA, Salisbury, Maryland
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I: Phase I: Patients receive oral SAHA twice daily on days 1-14 and bevacizumab IV over 30-90 minutes on day 1. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 6 patients are treated at the MTD.
  Phase II: Patients receive SAHA at the MTD determined in phase I and bevacizumab as in phase I.
  vorinostat: Given orally
  bevacizumab: Given IV
Period: Overall Study
Arm/Group | Arm I
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm I
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 64 [34 to 82]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Assessed by Response Evaluation Criteria for Solid Tumors (RECIST) (Phase II)
Description: Estimated by Kaplan-Meier method
Time Frame: At 6 months
Population: Progression free survival was summarized for the entire sample (n=37). The median survival times and 6-month survival rates are estim. based on the KP curve,w/ corresp. 95% confidence intervals using the log-log method. Conducted in SAS v9.3(Cary, NC). Progr.free survival time is calc. from date of first tx until date of progres./death or last fu.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Arm I
Number analyzed (Participants) | 37
percent | 48.6 [32 to 63.4]

2. Other Pre Specified Outcome: Maximum Tolerated Dose
Description: Determine the maximum tolerated dose of SAHA
Time Frame: 18 months from first patient dosing
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Clinical Response Rate of SAHA and Bevacizumab
Description: To determine the clinical response rate of SAHA and Bevacizumab in patients with metastatic renal cell carcinoma.
Time Frame: 7 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 7 years
Description: Adverse events were assessed through a regular investigator assessment
Arm/Group | Arm I
Serious Adverse Events (participants affected / at risk) | 3/37
Other Adverse Events (participants affected / at risk) | 22/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=37)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=37)
fatigue (Nervous system disorders) | 22 (22)
nausea (Gastrointestinal disorders) | 17 (17)
anorexia (Gastrointestinal disorders) | 16 (16)
diarrhea (Gastrointestinal disorders) | 13 (13)
elevated creatinine (Hepatobiliary disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less